CLINICAL TRIAL: NCT03789370
Title: Maintenance of Anaesthesia With Sevoflurane Versus Propofol and the Occurrence of Postoperative Headache.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Chrysanthi Batistaki, Assistant Professor of Anaesthesiology, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 06-11-14
Record Dates: First submitted 2018-01-15; First posted 2018-12-28 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the outcomes assessor will not know what kind of anaesthetic drug was used for maintainance of anaesthesia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol (Active Comparator): Total intravenous anaesthesia with propofol for maintainance of anaesthesia.Dose adjusted according to the Bispectral Index (BIS) indication (maintained 40-50). Initial dose 10 mg/kg/h for10 min, 8 mg/kg/h for 10 min and then 6 mg/kg/h).
  Interventions: Drug: Propofol
- Sevoflurane (Active Comparator): Sevoflurane for maintainance of anaesthesia. Dose 1 MAC adjusted according to the Bispectral Index (BIS) indication (maintained 40-50).
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Maintanance of general anaesthesia with propofol
  Arms: Propofol
Drug: Sevoflurane — Maintainance of general anaesthesia with sevoflurane.
  Arms: Sevoflurane

SUMMARY:
Postoperative headache is a major issue after general anaesthesia and surgery. The aim of this study is to investigate the possible difference in the occurrence of postoperative headache when general anaesthesia is maintained with propofol, which is supposed to have protective effects on migraine patients, versus sevoflurane.

DETAILED DESCRIPTION:
Postoperative headache is a major issue after general anaesthesia and surgery. The aim of this study is to investigate the possible difference in the occurrence of postoperative headache when general anaesthesia is maintained with propofol, versus sevoflurane. Propofol acts throught a GABA, and is known to have a therapeutic effect on migraine patients with accute attacts. However, its role on postoperative headache has not been studied, when used for maintainance of anaesthesia, this study aims to investigate the occurrence of headache after anaesthesia and surgery, when patients receive randomly two different anaesthetics: propofol and sevoflurane.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* scheduled operation under general anaesthesia
* operations <4 hours
* minorgynaecological operatios (leiomyomectomy)
* hernia repair
* arthroscopic procedurs
* minor orthopaedic operations without the use of tourniquet or cement
* saphenectomy
* minor urologic operations
* minor other operations of general surgery

Exclusion Criteria:

* age <18 and >65 years old
* ASA>III
* Diseases of the central nervous system (ie Parkinsons's disease, Multiple sclerosis, previous ischaemic attack, hydrocephalus, seizure disorder, etc)
* Psychosis under medication
* Cognitive impairement or/and inability to fill in the questionaires
* Allergy or contraindication to the study protocol included drugs
* Operations of more than 4 hours duration
* Head and neck procedures, procedures with neck extension (eg thyroidectomy), ENT procedures
* renal impairement
* hepatic impairement
* patient refusal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2014-11-07 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-10-30 (Estimated)

PRIMARY OUTCOMES:
incidence of postoperative headache (yes or no) | up to 24 hours postoperatively
  Rate of postoperative headache in patients receiving sevoflurane versus propofol (yes or no headache)

SECONDARY OUTCOMES:
Nausea and vomiting | up to 24 hours postoperatively
  Which anaesthetic (propofol or sevoflurane) is associated with less postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Anesthesiology, Attikon Hospital, 1 Rimini str., Athens, Greece